CLINICAL TRIAL: NCT07015307
Title: Study and Design of New Sustainable Exercise and Dietary-nutritional Programs for the Treatment of Metabolic Disorders in Elderly Women
Brief Title: Sustainable Exercise and Nutrition Programs for Managing Metabolic Disorders in Older Women
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alicante (Other)
Responsible Party: Principal Investigator, Prof. Dr. Alejandro Martínez-Rodríguez, Alejandro Martínez-Rodríguez, University of Alicante
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UA-2025-05-19_1
Record Dates: First submitted 2025-06-03; First posted 2025-06-11 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Metabolic Syndrome; Aging; Sarcopenia; Obesity; Chronic Disease; Frailty
Keywords: Mediterranean diet; Functional training; Women over 65; Lifestyle intervention; Nutrition and exercise
MeSH Terms: conditions — Metabolic Syndrome; Sarcopenia; Obesity; Chronic Disease; Frailty; Motor Activity

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to parallel intervention groups (dietary strategy, physical exercise, or combined). No crossover will occur between arms.
Who Masked: Outcomes Assessor
Masking Description: The researcher performing the statistical analysis will not know which intervention each group received.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Control - Healthy Women (No Intervention): Women over 65 years of age with no diagnosed metabolic alterations. Participants will follow their usual lifestyle without any specific nutritional or physical exercise intervention
- Control - Metabolic Alterations (No Intervention): Women over 65 years of age with metabolic alterations. Participants will continue their habitual routines without intervention, serving as a control group for comparison with the intervention arms.
- Diet Intervention (Experimental): Women with metabolic alterations will follow a sustainable dietary intervention based on Mediterranean principles. Personalized meal plans and regular follow-up will be delivered over a 12-week period. The aim is to improve metabolic and inflammatory markers.
  Interventions: Behavioral: Sustainable Diet Program
- Exercise Intervention (Experimental): Participants will perform a supervised physical exercise program focused on strength and functional training over 12 weeks. Exercises will be tailored to the participants' physical condition and delivered through structured sessions.
  Interventions: Behavioral: Supervised Physical Exercise Program
- Combined Diet + Exercise (Experimental): Participants will follow both the sustainable diet and the exercise program over a 12-week intervention period. This group will help assess the potential synergistic effect of the combined lifestyle strategies.
  Interventions: Behavioral: Combined Sustainable Diet and Exercise Program

INTERVENTIONS:
Behavioral: Sustainable Diet Program — Intervention based on the Mediterranean sustainable diet. It emphasizes the consumption of fish, fruits, and vegetables, while reducing the intake of meat and meat-derived products. The diet is tailored to the participants' health status, activity level, and nutritional requirements, following the recommendations of the Spanish Society of Cardiology and Endocrinology. Macronutrient and micronutrient goals follow national guidelines and are tracked using specialized dietary software.
  Arms: Diet Intervention
Behavioral: Supervised Physical Exercise Program — A 12-week supervised physical exercise program led by certified professionals in Sport Sciences. Exercise prescriptions are tailored individually based on baseline assessments and international guidelines from fields such as cardiology and metabolism. The sessions may include strength, endurance, or combined training. In the supervised period, the instructor guides the sessions, while during the unsupervised period, exercises are followed via an online platform that provides detailed explanations and graphics.
  Arms: Exercise Intervention
Behavioral: Combined Sustainable Diet and Exercise Program — This experimental arm combines the dietary intervention based on the sustainable Mediterranean diet with the structured physical exercise program. Both components are personalized and adhere to national and international health and nutrition recommendations. The program includes a 12-week supervised phase and an unsupervised online phase, aiming to maximize improvements in metabolic, physical, and psychosocial health in older women with metabolic alterations.
  Arms: Combined Diet + Exercise

SUMMARY:
This study aims to evaluate the impact of sustainable diet and exercise programs on metabolic health and quality of life in older women. Participants will be assigned to different intervention groups including supervised physical training, personalized dietary guidance based on the Mediterranean dietary pattern, or a combination of both. The programs will be implemented over several weeks, with continuous monitoring of variables such as body composition, functional capacity, strength, fatigue perception, sleep quality, and emotional well-being. The project also includes the development of a digital platform to support remote engagement and long-term health behavior change.

DETAILED DESCRIPTION:
This is a multi-phase interventional study designed to evaluate the impact of sustainable dietary and physical activity programs on metabolic health, functional capacity, and quality of life in older women. The target population includes women aged 65 and older, both with and without metabolic alterations.

The study comprises three phases:

Phase 1 includes initial assessments and an observational comparison between healthy older women and those with metabolic alterations.

Phase 2 implements three 12-week intervention programs: (1) a sustainable dietary strategy based on the Mediterranean diet, (2) a structured physical exercise program (both supervised and unsupervised), and (3) a combined intervention integrating both diet and exercise. Participants are assigned to groups based on their health status and intervention type.

Phase 3 focuses on knowledge transfer through the development of practical guidelines and a digital platform to facilitate remote monitoring and promote long-term adherence to healthy behaviors.

Primary and secondary outcomes include anthropometric measurements, body composition, handgrip strength, lower limb strength, walking speed, cardiovascular endurance, basal metabolic rate, blood pressure, blood biomarkers (glucose, cholesterol, triglycerides), fatigue perception, sleep quality, stress levels, emotional well-being, and health-related quality of life. Validated tools such as indirect calorimetry, digital hand dynamometers, functional capacity tests, and the SF-36 questionnaire will be employed.

The results are expected to support the design of sustainable, non-pharmacological strategies for the prevention and management of metabolic disorders and functional decline in aging women.

ELIGIBILITY:
Inclusion Criteria:

* Female participants aged 65 years or older
* Ability to walk independently or with assistive device
* Capacity to provide informed consent
* For groups with metabolic alterations: clinical diagnosis of metabolic syndrome based on standard criteria
* For healthy volunteers: absence of diagnosed metabolic or cardiovascular disease

Exclusion Criteria:

* Diagnosed cognitive impairment or dementia
* Unstable cardiovascular, respiratory, or musculoskeletal condition
* Participation in another structured lifestyle intervention during the study
* Any medical contraindication for physical exercise
* Severe mobility limitation preventing safe participation

Min Age: 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Gender Based: Yes — This study is exclusively for biologically female participants aged 65 and older due to its focus on aging-related metabolic changes in women.
Enrollment: 140 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Weight | Baseline (Week 0) and Week 12
  Measured in kilograms using a calibrated digital scale.
Heigth | Baseline (Week 0) and Week 12
  Measured in centimeters using a fixed wall-mounted stadiometer.
BMI | Baseline (Week 0) and Week 12
  Calculated as weight (kg) divided by height squared (m²), using measurements taken as above.
Waist circunference | Baseline (Week 0) and Week 12
  Measured in centimeters using a flexible, non-elastic anthropometric tape at the midpoint between the last rib and the iliac crest.
Body fat percentage | Baseline (Week 0) and Week 12
  Measured using multifrequency bioelectrical impedance.
Health-related quality of life (SF-36 score) | Baseline (Week 0) and Week 12
  Measured using the 36-Item Short Form Health Survey (SF-36), validated in Spanish (Vilagut, 2005), which assesses 8 domains of quality of life. Scores range from 0 to 100, with higher scores indicating better health-related quality of life.
Fatigue and perceived effort | Baseline (Week 0) and Week 12
  Measured with the Fatigue Severity Scale (FSS), a validated questionnaire that includes 9 items rated on a 7-point Likert scale. Scores range from 1 to 7, with higher scores indicating greater fatigue and perceived effort.
Energy intake (kcal/day) | Baseline (Week 0) and Week 12
  Total daily energy intake assessed through 3-day dietary records and a validated food frequency questionnaire for the Spanish population. Energy intake will be calculated in kilocalories per day (kcal/day) using standardized nutrient databases.
Carbohydrate intake | Baseline (Week 0) and Week 12
  Average daily carbohydrate intake measured through 3-day dietary records, expressed in grams. Higher values indicate greater carbohydrate consumption.
Protein intake | Baseline (Week 0) and Week 12
  Average daily protein intake measured through 3-day dietary records, expressed in grams. Higher values indicate greater protein consumption.
Fat intake | Baseline (Week 0) and Week 12
  Average daily fat intake measured through 3-day dietary records, expressed in grams. Higher values indicate greater fat consumption.
Daily step count | Baseline (Week 0) and Week 12
  Average number of steps per day measured with an accelerometer-based activity tracker. Higher scores indicate higher physical activity levels.
Active minutes per day | Baseline (Week 0) and Week 12
  Daily time spent in moderate to vigorous physical activity, measured in minutes per day using an accelerometer. Higher scores indicate higher physical activity levels.
Sedentary time per day | Baseline (Week 0) and Week 12
  Average number of minutes per day spent in sedentary behavior (e.g., sitting or lying down), measured via accelerometer. Higher scores indicate greater sedentary behavior (worse outcome).
Sleep quality (PSQI total score) | Baseline (Week 0) and Week 12
  Measured using the Pittsburgh Sleep Quality Index (PSQI), which provides a global score based on 19 items grouped into 7 components. Total scores range from 0 to 21, where higher scores indicate poorer sleep quality. PSQI score (range: 0-21).
Gait speed (10-meter walk test) | Baseline (Week 0) and Week 12
  Assessed by measuring the time to walk 10 meters at usual pace using infrared photocells (Chronojump, Barcelona, Spain).
Cardiovascular endurance (6-minute walk test) | Baseline (Week 0) and Week 12
  Evaluated using the 6-minute walk test (6MWT). Distance walked in 6 minutes on a flat surface, timed with a chronometer. Conducted on the athletics track at the University of Alicante.
Handgrip strength | Baseline (Week 0) and Week 12
  Measured using a digital hand dynamometer. Maximum isometric voluntary contraction recorded in the dominant hand.
Lower-limb isometric strength | Baseline (Week 0) and Week 12
  Assessed through maximum isometric voluntary contraction of the lower limbs using Kinvent force sensors and biofeedback platform.
Sarcopenia diagnosis | Baseline (Week 0) and Week 12
  Assessed according to the European Working Group on Sarcopenia in Older People criteria (EWGSOP, Cruz-Jentoft et al., 2010), using muscle strength, muscle mass and functional performance.
Basal metabolic rate | Baseline (Week 0) and Week 12
  Measured using indirect calorimetry
Systolic and diastolic blood pressure | Baseline (Week 0) and Week 12
  Assessed using an automatic digital sphygmomanometer (Omron Healthcare, Osaka, Japan), following standardized measurement protocol.
Cholesterol | Baseline (Week 0) and Week 12
  Measured using the Accutrend Plus analyzer (Roche Diagnostic, Mannheim, Germany) from capillary blood samples.
Triglycerides | Baseline (Week 0) and Week 12
  Measured using the Accutrend Plus analyzer (Roche Diagnostic, Mannheim, Germany) from capillary blood samples.
Glucose | Baseline (Week 0) and Week 12
  Measured using the Accutrend Plus analyzer (Roche Diagnostic, Mannheim, Germany) from capillary blood samples.

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Martínez Rodríguez, Dr., Principal Investigator — Alicante University
Locations (1):
- European Institute Of Exercise and Health, Elche, Alicante, Spain

IPD SHARING:
Plan to Share IPD: No